CLINICAL TRIAL: NCT04043442
Title: Neural Target Identification for Functional Disability Associated With Alcohol Related Characteristics Among Veterans With Co-occurring Alcohol Use Disorder and Traumatic Brain Injury
Brief Title: rTMS Target Identification for Functional Disability in AUD+mTBI
Acronym: rTMS-TARGET-ID
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2916-R; I01RX002916 (NIH)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder; Mild Traumatic Brain Injury
MeSH Terms: conditions — Alcoholism; Brain Concussion

STUDY DESIGN:
Intervention Model Description: Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P and Magpro C-B60
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Single Blind. A single blind will be maintained. Veterans will not know when they are receiving which treatment. Researchers will be unblinded to treatment order.
  rTMS Device and Blinding Procedures. PLACEBO and ACTIVE rTMS will be delivered with the Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P, which can be switched to active or placebo (A/P). The PLACEBO rTMS looks, sounds, and feels like ACTIVE rTMS. Each rTMS treater will be assigned a specific site of stimulation (Group 1, 2, 3, or 4) and will be blinded to the anatomical location of the other 3 sites. rTMS treaters and assessment administrators will be different people for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active + Placebo rTMS for Custom Neural Target Group 1 (Active Comparator): Custom neural anatomical target 1 defined by neuroimaging data
  Interventions: Device: Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P
- Active + Placebo rTMS for Custom Neural Target Group 2 (Active Comparator): Custom neural anatomical target 2 defined by neuroimaging data
  Interventions: Device: Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P
- Active + Placebo rTMS for Custom Neural Target Group 3 (Active Comparator): Custom neural anatomical target 3 defined by neuroimaging data
  Interventions: Device: Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P
- Active + Placebo rTMS for Left DLPFC Neural Target (Active Comparator): Neural anatomical target will be the Left Dorsolateral Prefrontal Cortex identified using the 5cm from the motor "hot spot" rule.
  Interventions: Device: Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P

INTERVENTIONS:
Device: Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P — rTMS device
  Other Names: rTMS device

SUMMARY:
The objectives of this VA Merit application are to identify a neural target unique to Veterans with co-occurring alcohol use disorder and mild traumatic brain injury (AUD+mTBI) and to test the efficacy of this target as a stimulation site for repetitive transcranial magnetic stimulation (rTMS) treatment to maximize functional recovery. rTMS will soon be a treatment option at 30 VAs nationwide and preliminary studies show promise for AUD and mTBI treatment. A better understanding of how AUD+mTBI impacts the brain needs to occur in order to advance rTMS to optimize function. This research is aligned with the VA RR&D's mission to generate knowledge and innovations to advance the rehabilitative health and care of Veterans, to effectively integrate clinical and applied rehabilitation research, and translate research results into practice. This research is also aligned with the goal of the Psychological Health & Social Reintegration portfolio to develop interventions improving psychological health status of Veterans enabling them to function more fully in society.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) and mild traumatic brain injury (mTBI) impact functional abilities. AUD occurs in up to 35% of Veterans with mTBI. Evidence suggests that co-occurrence of AUD and mTBI (AUD+mTBI) leads to an exacerbation of brain dysfunction, symptom manifestation, and ultimately, functional disability. Alcohol-related characteristics are operationally defined per AUD symptoms and outcomes including, but not limited to, alcohol consumption, alcohol craving, and AUD severity. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulatory treatment that will soon be a treatment option at 30 VAs nationwide. Preliminary rTMS efficacy is demonstrated for AUD alone and mTBI alone using a variety of neural targets. rTMS is, thus, a promising treatment for AUD+mTBI. The objectives of this study are to 1) identify neural targets (i.e. site of stimulation) associated with both alcohol-related characteristics and self-reported functional disability, and 2) assess preliminary efficacy and sustainability of a high frequency rTMS protocol applied to these customized neural targets relative to the commonly used left dorsolateral prefrontal cortex (DLPFC) site. Addressing these objectives are essential steps towards the long-term research goal [to customize and clinically implement a rTMS treatment] that can improve brain function resulting in optimal recovery for Veterans with AUD+mTBI. To address the first study objective, Veterans will be recruited and classified into one of two groups based on structured-interviews, self-report measures, and neuropsychological assessments: 1) AUD+mTBI, and 2) [Veteran controls] without a history or symptoms of mTBI or AUD. Alcohol-related characteristics will be assessed through objective measures of alcohol use, self-report measures, and structured interviews. Self-reported functional disability will be assessed using the World Health Organization Disability Assessment Schedule 2.0 (WHODAS). Neuroimaging metrics will be assessed through a multi-modal, functional and structural Magnetic Resonance Imaging (MRI) scan. Participants will complete a functional MRI (fMRI) protocol where brain activation will be measured in response to viewing images related to alcohol, compared to neutral images. Advanced neuroimaging procedures to determine the structural integrity of white matter fibers in the brain and spontaneous activity in brain networks, a process called resting state functional connectivity (rsFC), will also be conducted. To address the second study objective, AUD+mTBI Veterans will receive rTMS at one site randomly assigned from a set of 4 sites: 3 customized neural targets identified in this study, and the commonly used left DLPFC. AUD+mTBI Veterans will complete 10 PLACEBO, then 10 ACTIVE rTMS sessions in a within-subjects design. Follow-up WHODAS assessments will occur at 2-weeks, 1-month and 6-months post-ACTIVE rTMS. Aim 1 will identify unique neural targets for rTMS to treat AUD+mTBI by determining which multi-modal neuroimaging metrics are most strongly associated with both alcohol-related characteristics and functional disability. Aim 2 will [test preliminary efficacy of high-frequency rTMS administered over the customized neural targets] to treat functional disability among Veterans with AUD+mTBI. Aim 3 will assess sustainability of rTMS effects on functional disability for Veterans with AUD+mTBI. The investigators hypothesize that for Veterans with AUD+mTBI, there are neural substrates of AUD related to functional disability, and that neuromodulation of these substrates will be related to gains in functional disability. The investigators' innovative approach represents an advancement in the field of neurorehabilitation because a neural target will be systematically defined, using multi-modal neuroimaging, prior to preliminary rTMS efficacy and sustainability testing. These steps are necessary to customize rTMS treatment for a population of Veterans with co-occurring conditions and unique health care needs. Thus, the outcomes of this research will optimize function for Veterans with AUD+mTBI.

ELIGIBILITY:
Inclusion Criteria:

* Can read and speak English
* Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for AUD
* Symptom Attribution and Classification (SACA) criteria (Pape, Herrold et al 2016, JHTR) for mTBI (without requirement of clinical neuropsychological impairment)

Exclusion Criteria:

* History of moderate to severe TBI
* Neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease, multiple sclerosis)
* History of or current psychotic spectrum disorders (i.e., schizophrenia, schizoaffective and bipolar disorders)
* Intellectual disability (WTAR predicted full-scale IQ score < 70)42
* Are pregnant or nursing
* Use of benzodiazepines, opiates, cocaine, or amphetamines in the past 30 days
* Meet DSM-5 criteria for moderate to severe cannabis use disorder
* Contraindications to MRI (e.g., claustrophobia, ferromagnetic metal in eyes or face, congestive heart failure, implanted cardiac pacemaker or defibrillator, cochlear implant, nerve stimulator)
* Meet SACA criteria for 'Questionable Validity' of performance effort and symptom reporting

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) Change | baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 6 months
  36-item self report measure of global functional disability. We will use the complex scoring method which creates a summary score into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability).

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Herrold, PhD BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. MRI images will anonymized and made available through the Northwestern University Neuroimaging Data Archive (NUNDA). Final data sets will be made available as per Hines VA Hospital local policy for long term storage and access until enterprise-level resources become available. These data will be available upon request by researchers and scientists in accordance with federal guidelines and Hines local policy.The data provided will be sufficient for anyone to perform analogous or supplemental analyses that would permit validation of the analysis and results. The sharing of data will enable others to evaluate the data and to validate and interpret the data independently. In order to insure that replication is possible and transparency, statistical code complementary to datasets will be made available through the Federal Interagency Traumatic Brain Injury Research Informatics System.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Three years after study completion or after all primary papers have been accepted for publication.
Access Criteria: Federal Interagency Traumatic Brain Injury Research Informatics System.

REFERENCES:
- [Derived] Herrold AA, Aaronson AL, Bhaumik D, Durazzo T, Livengood SL, Ramic A, Riordan P, Jordan N, Parrish T, Mallinson T, Kale IO, Billups A, Krese K, Kletzel S, Philip NS, Bender Pape TL. A Customized Neural Transcranial Magnetic Stimulation Target for Functional Disability Among Veterans With Co-Occurring Alcohol Use Disorder and Mild Traumatic Brain Injury: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 23;14:e64909. doi: 10.2196/64909. PMID 40550124